CLINICAL TRIAL: NCT07169981
Title: Effect of Empagliflozin 10 vs 25 mg on LV Remodeling in Diabetic Patients With Anterior STEMI With Reduced LVEF Who Underwent Primary PCI
Brief Title: Effect of Empagliflozin 10 vs 25 mg on LV Remodeling in Diabetic Patients With Anterior STEMI With Reduced LVEF
Acronym: EMPA-DMMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD 100/2023
Record Dates: First submitted 2025-08-20; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-07

CONDITIONS: Diabete Mellitus; Heart Failure; Remodeling, Left Ventricle
Keywords: Empagliflozin; Heart Failure; Left Ventricular Remodeling; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure; Ventricular Remodeling | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin 10 mg (Experimental): Participants in this arm will receive Empagliflozin 10 mg orally once daily for a duration of 6 months. The purpose is to evaluate the effect of Empagliflozin on left ventricular remodeling and cardiac function in patients with HFrEF. Standard heart failure therapy may be continued alongside the study drug as clinically indicated.
  Interventions: Drug: Empagliflozin 10 MG [Jardiance]
- Empagliflozin 25 mg (Experimental): Participants in this arm will receive Empagliflozin 25 mg orally once daily for a duration of 6 months. The purpose is to evaluate the effect of Empagliflozin on left ventricular remodeling and cardiac function in patients with HFrEF. Standard heart failure therapy may be continued alongside the study drug as clinically indicated.
  Interventions: Drug: empagliflozin (Jardiance) 25 mg

INTERVENTIONS:
Drug: Empagliflozin 10 MG [Jardiance] — This intervention consists of Empagliflozin 10 mg oral tablets administered once daily for a duration of 6 months. The drug is used in this study to evaluate its effect on left ventricular remodeling in patients with heart failure. Empagliflozin is a sodium-glucose co-transporter 2 (SGLT2) inhibitor approved for the treatment of type 2 diabetes and heart failure. In this trial, it is being investigated specifically for its impact on cardiac structure and function.
  Arms: Empagliflozin 10 mg
Drug: empagliflozin (Jardiance) 25 mg — This intervention consists of Empagliflozin 25 mg oral tablets administered once daily for a duration of 6 months. The drug is used in this study to evaluate its effect on left ventricular remodeling in patients with heart failure. Empagliflozin is a sodium-glucose co-transporter 2 (SGLT2) inhibitor approved for the treatment of type 2 diabetes and heart failure. In this trial, it is being investigated specifically for its impact on cardiac structure and function.
  Arms: Empagliflozin 25 mg

SUMMARY:
This study is investigating how the medication Empagliflozin affects the heart's structure and function in patients with heart disease. Empagliflozin is already used to treat diabetes and heart conditions, and this research aims to see if it can help improve heart remodeling, which may lead to better heart health and quality of life. Participants will receive the medication and have regular check-ups to monitor their progress. The study is carefully designed to ensure participant safety. If you have heart disease and want to learn more, please contact (hany_barsoum@med.asu.edu.eg).

DETAILED DESCRIPTION:
Heart disease is a leading cause of illness worldwide, and new treatments that improve heart function can have a significant impact on patient health and longevity. This research could provide valuable insights into how existing medications can be used to benefit people with heart conditions beyond their current use.

This clinical study aims to understand how Empagliflozin, a medication commonly used to treat diabetes, affects the heart's structure and function in people with heart disease. When the heart is damaged, especially on the left side (left ventricle), it can change shape and size-a process called remodeling-which may reduce how well the heart pumps blood. This study will explore whether Empagliflozin can help reverse or improve this remodeling process, potentially leading to better heart function and improved quality of life.

Participants in the study will receive Empagliflozin and undergo regular health check-ups, including imaging tests like echocardiograms, to track changes in heart structure and performance. The study is designed to carefully monitor safety and effectiveness, ensuring participants are supported throughout.

If you or a loved one has heart disease and are interested in learning more about this study, please contact [hany_barsoum@med.asu.edu.eg].

ELIGIBILITY:
Inclusion Criteria:

Diabetic patients with anterior STEMI with reduced LVEF who underwent PPCI with successful revascularization and resulting into TIMI III flow and who are receiving SGLTi for the first time.

Exclusion Criteria:

1. patients who did not undergo primary PCI, those treated medically or had thrombolysis
2. Non diabetic patient.
3. Diabetic patient already on SGLTi
4. STEMIs other than anterior.
5. NSTEMI patients.
6. Patients having valvular heart diseases.
7. Patients having renal impairment.
8. Patients with LV myopathies of non-ischemic origin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
left ventricular remodeling | 6 months
  change of left ventricular volumes form baseline and after 6 months
left ventricular systolic function | 6 months
  change of left ventricular ejection fraction from baseline and after 6 months
left ventricular Global Longitudinal Strain (GLS) | 6 months
  changes of GLS from baseline and after 6 months

SECONDARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | 6 months
  MACE is defined as a composite of cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke.
Assessment of diastolic function | 6 months
  studying the effect of different doses of Empagliflozin not only on systolic function but also on diastolic function with E/E'
Left Atrial Strain | 6 months
  studying the effect of different doses of Empagliflozin on Left Atrial Strain

CONTACTS AND LOCATIONS:
Overall Officials: Zainab A. Fahmy, Professor of Cardiology, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT07169981/Prot_000.pdf